CLINICAL TRIAL: NCT01855932
Title: Enlighten: An Adaptive Technology Weight Loss Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Bonnie Spring, Principal Investigator, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: STU00078810
Record Dates: First submitted 2013-05-10; First posted 2013-05-17 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2013-09

CONDITIONS: Obesity; Weight Loss
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Technology Supported (Experimental)
  Interventions: Behavioral: Technology Supported

INTERVENTIONS:
Behavioral: Technology Supported — All participants will complete 8 weeks of recording of dietary intake, weight, and physical activity on a smartphone application. Time-stamped data from the smartphone will upload automatically to the application server, where it will be visible to the lifestyle coach. The participant's real-time diet, activity and weight data relative to their goals will be visually depicted on the participant's smartphone. The coach will monitor participant adherence and send supportive text messages. Response to the application will be assessed 3 weeks after enrollment into the study; measured by number of food items recorded between weeks 1-3 of the intervention; an indicator of use and adherence. Based on adherence, some participants may receive 4 telephone coaching sessions between weeks 5 and 8. Telephone coaching sessions will include feedback on self-monitoring and goal attainment, problem solving, and motivational interviewing.

SUMMARY:
The Enlighten study is an 8-week trial investigating the response to use of a smartphone diet and activity application. Participants are enrolled as part of a worksite intervention, and will receive the LoseIt! weight loss smartphone application, which requires participants to self-monitor dietary intake and physical activity, a component shown to effectively produce weight loss. The application will be programmed to deliver dietary intake recommendations during the first three weeks of the intervention. At the 3 week time point, self-monitoring adherence via the smartphone application will be assessed and those who are not responding will receive 4 weekly telephone coaching sessions. Those individuals who respond at the end of 3 weeks will be encouraged to continue self-monitoring on the application. All participants will also receive regular text messages throughout the trial. The importance of the proposed research lies in the objective to reconfigure weight loss treatment so as to achieve the intended outcome more efficiently and in a manner that allows greater reach.

ELIGIBILITY:
Inclusion Criteria:

* BMI greater than 25-39.9 kg/m2
* Weigh no more than 300 pounds.
* Weight stable (no loss or gain >25 lbs for the past 6 months)
* Not enrolled in any formal weight loss program
* Not currently taking anti-obesity medications
* Interested in losing weight
* Own an Android Smartphone or iPhone, be willing to install the Lose It! Application, and agree to join the Enlighten group which will allow study staff to view participant data using a private coaching interface.

Exclusion Criteria:

* Unstable medical conditions (uncontrolled hypertension, diabetes, unstable angina pectoris, myocardial infarction, transient ischemic attack, cancer undergoing active treatment, or cerebrovascular accident within the past six months)
* History of diabetes requiring insulin supplementation
* Crohn's Disease
* Diagnosis of obstructive sleep apnea requiring intervention (i.e. CPAP)
* Require use of an assistive device for mobility (e.g., wheelchair, walker, cane)
* BMI greater than or equal to 40, weight greater than or equal to 300 pounds
* Hospitalization for a psychiatric disorder within the past 5 years
* Those at risk for adverse cardiovascular (CVD) events with moderate intensity activity
* Those who cannot read the study questionnaires will be excluded
* Those currently taking weight loss medication or committed to following an incompatible dietary regimen.
* Female participants may not be pregnant, trying to get pregnant, or lactating.
* Bulimia Nervosa
* Binge Eating Disorder
* Active Suicidal Ideation
* those on medications known to cause weight gain (e.g., prednisone)
* current substance abuse or dependence besides nicotine dependence
* low motivation to change that would interfere with program adherence

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-05; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change in Anthropometric Measures | Baseline, 8 Weeks
  Weight, Waist Circumference, Blood Pressure
Self-Monitoring Adherence over Time | Baseline, 8 weeks
  Diet,Activity & Weight Self-Monitoring

SECONDARY OUTCOMES:
Demographics | Baseline
Call Session Adherence | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie J Spring, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States